CLINICAL TRIAL: NCT05867355
Title: A Multi-Centre Prospective Cohort Study of Surgically Treated Displaced Mid-diaphyseal Clavicle Fractures
Brief Title: Surgically Treated Displaced Mid-diaphyseal Clavicle Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Unity Health Toronto (Other); Winnipeg Regional Health Authority (Other); Thunder Bay Regional Health Sciences Centre (Other); Montreal General Hospital (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Prism Schneider, Orthopedic Trauma Research Lead, University of Calgary
Other Study IDs: REB20-2049
Record Dates: First submitted 2023-05-04; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Clavicle Fracture
MeSH Terms: interventions — Surgical Fixation Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical fixation — compare implant removal rates between surgical fixation techniques.

SUMMARY:
This prospective, multi-centre study aims to determine clinical, radiographic, and patient-reported outcomes (PROMs) following surgical fixation of displaced mid-diaphyseal clavicle fractures and to compare implant removal rates between techniques within 2-years of the procedure.

DETAILED DESCRIPTION:
Given the substantially lower implant removal rate in combination with a high union rate with the dual mini-fragment technique, we do not believe there is clinical equipoise required for a randomized clinical trial.

This study is a multi-centre, prospective cohort study (11 sites confirmed to date) of all operatively treated clavicle fractures, in order to objectively evaluate all current surgical techniques used across Canada. This pragmatic approach will allow us to observe surgical decision-making, rationale for implant removal, and report on clinical, radiographic, and patient-reported outcomes for all techniques over a 2-year follow-up timeframe, for the first time.

All enrolled patients will be encouraged to begin immediate range of motion as tolerated and weightbearing as tolerated post-operatively. This will be assessed at each follow-up and any reason for delayed motion or weightbearing will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Treated with surgical fixation for a displace mid-diaphyseal clavicle fracture.
* Aged 18 years of age or older and skeletally mature.
* Enrolled within 21 (+3 days) of injury.
* Willing and able to complete consent and study participation.

Exclusion Criteria:

* Pathological fractures.
* Clavicle non-unions.
* Current or prior ipsilateral upper extremity injury that may impact functional outcomes.
* Polytrauma patients with injuries projected to affect rehabilitation course.
* Active malignancy.
* Inability to provide consent or complete follow-up.
* Incarcerated patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Skeletally mature, adult participants aged 18 years of age or older, who are treated with surgical fixation for a displaced mid-diaphyseal clavicle fracture. Exclusion criteria: Pathological fractures, clavicle non-unions, current or prior ipsilateral upper extremity injury that may impact functional outcomes, or an inability to consent or complete follow-up.
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine implant removal rates | 4 years
  To report implant removal rates in an appropriately powered prospective cohort study.
Identify rationale for implant removal | 4 years
  To report rationale for implant removal in an appropriately powered prospective cohort study.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada